CLINICAL TRIAL: NCT06943352
Title: Effects of Interactive Sensory Play on Manual Dexterity in Down Syndrome Children
Brief Title: Effects of Interactive Sensory Play on Manual Dexterity in Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/taiba hussain
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
Keywords: Interactive Sensory play; Manual Dexterity; Free Play
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be performed. Participants of this group will play in a group with sensory bins with other children. The intervention will help children interact with others in society and for improving manual dexterity. According to FITT Principle, the intervention will be given 3 days a week for 12 weeks and alternate days will be selected. After every 2 weeks, the tasks will be upgraded. The free play will be given for 15 minutes and interactive sensory play will be given for 30 minutes. The interventions will be given for 45 minutes in each session.
  Drawing and painting are involved in free play. Participants of group will play alone. The participants will draw or paint for improving manual dexterity. According to FITT Principle, the intervention will be given 3 days a week for 12 weeks and alternate days will be selected. After every 2 weeks, the tasks will be upgraded. The interventions will be given for 45 minutes in each session.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Sensory play with Free Play Group (Experimental): Participants of this group will play in a group with sensory bins with other children. The sensory bin is a basket filled with different objects of different shapes, sizes, and textures. The intervention will help children interact with others in society and for improving manual dexterity. The children play in group and alone also for this group.
  According to FITT Principle, the intervention will be given 3 days a week for 12 weeks and alternate days will be selected. At first, small and easy tasks will be given and after every 2 weeks, the tasks will be upgraded. The free play will be given for 15 minutes and interactive sensory play will be given for 30 minutes. The interventions will be given for 45 minutes in each session.
  Interventions: Other: Sensory Bins; Other: Drawing and Painting
- Free Play Group (Active Comparator): Drawing and painting are involved in free play. Participants of this group will play alone. The participants will draw or paint for improving manual dexterity. According to the FITT Principle, the intervention will be given 3 days a week for 12 weeks and alternate days will be selected. At first, small and easy tasks will be given and after every 2 weeks, the tasks will be upgraded. The interventions will be given for 45 minutes in each session.
  Interventions: Other: Drawing and Painting

INTERVENTIONS:
Other: Sensory Bins — The sensory bin is a basket filled with different objects of different shapes, sizes, and textures.
  Arms: Interactive Sensory play with Free Play Group
Other: Drawing and Painting — Colored pencils and watercolors will be used.

SUMMARY:
Down Syndrome is a genetic condition in which a patient has an extra chromosome which is a copy of chromosome 21. It causes physical, cognitive, and behavioral symptoms. The person has difficulty with normal life activities. This study evaluates the effect of interactive sensory play on coordinated hand movements or manual dexterity in children with Down Syndrome. Down syndrome is one of the most common birth defects and causes impairments in the body. The children diagnosed with Down syndrome need great deal of therapies in early childhood so that can live a better life. The objective of this study is to assess the effects of interactive sensory play on manual dexterity in Down syndrome children.

The study design will be a Randomized Controlled Trial. The study setting will be Tehsil Headquater hospital Sadiqabad. The study duration will be 10 months after the approval of the synopsis. The Sample Size will be 22 which is calculated by epitools. The sampling technique will be a Non-probability convenient sampling technique. Children who are diagnosed with Down Syndrome will be included. Children with other musculoskeletal and neurological issues will be excluded. Data Collection Tools will be Box and Block test and Pediatric Evaluation of Disability Inventory. Identification and recruitment of the participants with Down syndrome will be done. Participants will be selected through lottery for both groups. Group 1 will use Interactive Sensory play and Group 2 will use Free Play as intervention. The assessor will be blind. The data will be analyzed using SPSS 23.

ELIGIBILITY:
Inclusion Criteria:

* Children with moderate level of mental retardation who are able to follow commands

Exclusion Criteria:

* • Children with other musculoskeletal and neurological issues.

  * Children with down syndrome but also have complications such as epilepsy, congenital heart condition.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Box and Block test | At the start as baseline data. Again at 6th week and then finally at 12th week.
  This test is used to measure manual dexterity. This test is simple, cheap and quick. The test can be used for different populations to assess the coordinated movements of the hands. The test-retest reliability on more weak hand is 0.98 and the less weak hand is 0.93.It has good convergent validity as the value is 0.80.
• Pediatric Evaluation of Disability Inventory | At the start as baseline data. Again at 6th week and then finally at 12th week.
  This is an interviewing tool to assess the independence of the patients to perform different activities using their hands. The reliability that was seen was ranging from 0.18 to 0.94. The value of construct validity was seen to be ranging from 0.64-0.95.
Nine-Hole Peg Test | At the start as baseline data. Again at 6th week and then finally at 12th week.
  This test is used to assess manual dexterity. This test is easy, simple and quick. This test assess coordinated movements of hands. This test consists of a board with nine holes and square boxes or pegs which are inserted into the holes by the participants. This test can be used for assessment in every population. It has excellent interrater reliability which is equal to 0.75 to 0.99. It has excellent convergent validity that is equal to 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Taiba Hussain, MS-PPT, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jarusriboonchai P, Meissner JL, Almeida T, Balaam M. Understanding children's free play in primary schools. InProceedings of the 9th International Conference on Communities & Technologies-Transforming Communities 2019 Jun 3 (pp. 178-188).